CLINICAL TRIAL: NCT02210130
Title: Measure of Specific Determinants of the Cerebral Small Vessel Disease in HIV+ Patients
Brief Title: The Microvascular Brain Retina And Kidney Study
Acronym: MICROBREAK2
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Collaborators: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Other Study IDs: AMR_2013-8
Record Dates: First submitted 2014-08-05; First posted 2014-08-06 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Cerebral Small Vessels Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- patients HIV+ CSVD+: patients with HIV and cerebral small vessel disease
- control HIV+ CSVD-: patients with HIV and without cerebral small vessel disease

SUMMARY:
Cerebral small vessel disease (CSVD) is a major cause of cognitive impairment and disability in the general population, secondary to the accumulation of asymptomatic elementary lesions. CSVD is directly correlated with age and cardiovascular risk factors and therefore would be challenging in term of public health care in the future. While HIV patients share the same cardiovascular risk factors and they are often diagnosed with cognitive impairment and frailty, CSVD has not been yet described in this population.

The global aim is to study and describe the CSVD in the HIV+ population by: (1) correlating the CSVD and the macro-vascular disease of the head and brain; (2) correlating the CSVD with the ocular (structural sentinel organ) and kidney (functional sentinel organ) micro-vascular disease.

HIV+/CSVD+ patients will have a complementary work-up with conventional MRI/MRA, thorough vascular explorations, and neurologic examination to evaluate the severity of the CSVD, the macro-vascular disease and the cerebral atrophy. They will have a full ophthalmic examination and specific kidney explorations to evaluate the micro-vascular disease of this two sentinel organs. The same number of HIV+/CSVD- matched patients will have the same work-up.

We are expecting to show the relationship between CSVD and cardiovascular risk factors in order to propose specific prevention. We will correlate the CSVD with the neurologic and cognitive function as it is already proved in the general population. We will correlate the CSVD with the ocular and kidney micro-vascular disease to propose fast, easy and cheap screening tools for the CSVD in the HIV+ population.

ELIGIBILITY:
Inclusion Criteria:

* age over 50 years old
* chronic HIV seropositive patient infected for at least 5 years
* antiretroviral therapy
* plasmatic HIV viral load <40 copies/ml for at least one year with one authorized blip < 1000 copies/ml per year
* cerebral small vessels disease (patients) or not (controls)

Exclusion Criteria:

* Co-infection VHC
* known antecedent of stroke
* documented neurologic complication of HIV
* drug user
* glomerular filtration rate< 15 mL/mn
* diabetic patient with kidney or retin complications
* systolic blood pressure≥ 180 and/or diastolic blood pressure≥ 110 mmHg

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV patients over 50 years old, infected for at least 5 years, treated with antiretroviral (ARV) therapy With (patients) or without Cerebral Small Vessels Disease
Sampling Method: Non-Probability Sample
Enrollment: 163 (Actual)
Dates: Start 2014-05; Primary Completion 2014-05 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
determinants of CSCV in patients with HIV | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Ophtalmologique Adolphe de Rothschild, Paris, Île-de-France Region, France

REFERENCES:
- [Derived] Januel E, Godin O, Moulignier A, Lescure FX, Savatovsky J, Lamirel C, Valin N, Tubiana R, Canestri A, Roux P, Sadik JC, Salomon L, Katlama C, Yazdanpanah Y, Pialoux G, Girard PM, Costagliola D, Assoumou L; Microvascular Brain Retina And Kidney (MicroBREAK) Study Group. Brief Report: Impact of ART Classes on the Increasing Risk of Cerebral Small-Vessel Disease in Middle-Aged, Well-Controlled, cART-Treated, HIV-Infected Individuals. J Acquir Immune Defic Syndr. 2019 Aug 15;81(5):547-551. doi: 10.1097/QAI.0000000000002084. PMID 31107300